CLINICAL TRIAL: NCT06872788
Title: Study of Sensory Attenuation in Functional Movement Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aditya Murgai, Assistant Professot, Western University, Canada
Other Study IDs: 126375
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Functional Movement Disorder
Keywords: functional movement disorder; sensory attenuation; sense of agency
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Functional Movement Disorder
- Controls: Healthy subjects

SUMMARY:
Functional movement disorders (FMD) are conditions where people experience unusual movements or difficulties with walking, not caused by a specific brain or nerve injury but related to how the brain controls movements. Functional movement disorders are common in clinical practice and can lead to significant disability and healthcare costs.

A key feature of FMD is a problem with self-agency-the feeling that we are in control of our own movements. Many patients with FMD feel that their abnormal movements happen without their control. Sensory attenuation is closely linked to self-agency. It's the brain's way of reducing the intensity of sensations caused by our own movements. For example, you can't tickle yourself because your brain knows it's your own action. In people with FMD, this process doesn't work properly. As a result, they might feel their movements are involuntary.

Previous research shows that sensory attenuation is reduced in FMD, but the studies so far have been small. This study will investigate sensory attenuation in a larger group of FMD patients and compare it with healthy individuals. The goal is to see if reduced sensory attenuation could be used as a marker to measure the severity of FMD.

DETAILED DESCRIPTION:
Objective: The primary objective of the study is to investigate sensory attenuation in patients with functional movement disorders using the force-matching paradigm. The secondary objective is to determine whether sensory attenuation metrics are correlated with disability and functional movement disorder scores.

Materials: The data will be collected using a stand-alone, mechatronic system, capable of applying precise forces to a patient's finger and capturing a patient's force inputs into the system. This device has an integrated data collection system that ensures all results are captured and stored on an SD card.

Experimental Design: Thirty-five patients diagnosed with FMD and 35 healthy controls will be included in the study. Patients will be enrolled from the integrated functional movement disorders clinic and the movement disorders clinic at the London Health Sciences Center.

Each participant will be tested on two conditions: (1) Self condition: matching a target force by pressing on a movement arm with an integrated pressure transducer over the non-dominant index finger. (2) External condition: Matching a target force by moving a slider that controls the pressure generated by the movement arm placed over the non-dominant index finger. Five different target forces, with 0.5 Newtons increments, from 1 Newton to 3 Newtons, will be randomly presented in both conditions. All subjects will complete a total of 30 randomly generated forces for each condition. The applied forces are small and not painful.

Procedure: Participants will sit in front of a table and place the tip of their non-dominant index finger under the force transducer. In the self-condition (condition 1), the motor will exert one of the five target forces in each trial. The participants will then start matching the target force by directly pressing onto the movement arm, which rests on the non-dominant index finger, using the contralateral index finger. In the external condition (condition 2), the motor will exert one of the five target forces. The participant will then match the target force by moving a potentiometer slider, which controls the force generated by the movement arm placed over the non-dominant index finger. The study visit will be completed in one hour.

The ratio between the matched force and the target force will be calculated and serve as a sensory attenuation measure. This measure will be averaged across trials to give the mean attenuation for each force level and condition.

Statistical analysis: A Mixed Design ANOVA will be used to measure the differences between the within-subjects factors (conditions and force levels) and the between-subjects factor (healthy control vs. FMD groups). Post-hoc analysis will be conducted using Bonferroni correction for multiple comparisons to determine which specific means are significantly different. Pearson's correlation will be used to determine how scores on the World Health Organization Disability Assessment Schedule (WHODAS2) and the Psychogenic Movement Disorders Scale (PMDS) are related to the degree of sensory attenuation.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosed with a functional movement disorder (2) Age >18 years

Exclusion Criteria:

(1) Moderate to severe action tremor in the dominant hand that interferes with the tasks. (2) Upper limb peripheral neuropathy. (3) Inability to read or understand English.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: movement disorder clinic
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sensory attenuation measurement | Day 1
  The primary outcome of this study is to measure sensory attenuation in patients with functional movement disorders (FMD) using the force-matching paradigm. Sensory attenuation will be quantified by calculating the ratio of matched forces to target forces in both self and external conditions.

SECONDARY OUTCOMES:
Correlation between WHODAS2 and PMDS with sensory attenuation. | Day 1
  Correlation between The World Health Organization Disability Assessment Schedule (WHODAS2) and Psychogenic Movement Disorders scale (PMDS) scores with the amount of sensory attenuation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
At this time, IPD will not be shared due to confidentiality concerns.